CLINICAL TRIAL: NCT06069895
Title: Investigation of Safety, Tolerability and Pharmacokinetics of Multiple Doses of NNC0113-6856 in Healthy Participants, Including a Subset of Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9904-5008; U1111-1284-5743 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0113-6856 (Experimental): Participants will receive NNC0113-6856 oral tablets.
  Interventions: Drug: NNC0113-6856
- Placebo (Experimental): Participants will receive NNC0113-6856 matching placebo oral tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0113-6856 — NNC0113-6856 will be administered as oral tablets.
  Arms: NNC0113-6856
Drug: Placebo — NNC0113-6856 matching placebo will be administered as oral tablets.
  Arms: Placebo

SUMMARY:
NNC0113-6856 is a new medicine which may help participants with type 2 diabetes to improve blood sugar control. NNC0113-6856 is slowly converted in the body to semaglutide, a substance similar to a hormone (signaling substance) in the body. The main purpose of this study will be to evaluate the safety of different strengths of NNC0113-6856 when given as multiple administrations, and the amount of NNC0113-6856 in the blood will be measured as well as the amount of specific parts (including semaglutide). Participants will either get multiple doses of the new medicine NNC0113-6856 or multiple doses of placebo (a "dummy" medicine that looks like the new medicine but is without any active ingredient). Whether participants get the new medicine or placebo is decided by chance. The duration of the study could last up to 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 21.0 and 29.9 kilograms per meter square (kg/m^2) (both inclusive) at screening.

Additional for healthy Japanese participants:

* First generation Japanese (Japanese born participants).

Exclusion Criteria:

* HbA1c greater than or equal to (≥) 6.5 percent (%) (48 millimoles per mole [mmol/mol]) at screening.
* Any of the below laboratory safety parameters at screening outside the below laboratory range, see "Log of laboratory ranges used for laboratory parameter exclusion criterion" for specific values:

  1. Alanine Aminotransferase (ALT) greater than (>) upper normal limit (UNL) +10%
  2. Aspartate aminotransferase (AST) > UNL+20%
  3. Total bilirubin > UNL+20%
  4. Creatinine > UNL+10%
  5. International normalised ratio (INR) > UNL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | From time of first dosing (day 1) until completion of the follow-up visit (day 148)
  Measured as number of events.

SECONDARY OUTCOMES:
Part 1 Multiple ascending dose (MAD): AUCτ,sema,SS: area under the semaglutide plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in hours*nanomoles per liter (h*nmol/L).
Part 1 (MAD): Cmax,sema,SS: maximum observed plasma concentration of semaglutide at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nanomoles per liter(nmol/L).
Part 1 (MAD): AUCτ,6856,SS: area under the NNC0113-6856 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in h*nmol/L.
Part 1 (MAD): Cmax,6856,SS: maximum observed plasma concentration of NNC0113-6856 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nmol/L.
Part 1 (MAD): AUCτ,4768,SS: area under the NNC0113-4768 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in h*nmol/L.
Part 1 (MAD): Cmax,4768,SS: maximum observed plasma concentration of NNC0113-4768 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nmol/L.
Part 2 Dosing condition (DC): AUCτ,sema,SS: area under the semaglutide plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in h*nmol/L.
Part 2 (DC): Cmax,sema,SS: maximum observed plasma concentration of semaglutide at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in nmol/L.
Part 2 (DC): AUCτ,6856,SS: area under the NNC0113-6856 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in h*nmol/L.
Part 2 (DC): Cmax,6856,SS: maximum observed plasma concentration of NNC0113-6856 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in nmol/L.
Part 2 (DC): AUCτ,4768,SS: area under the NNC0113-4768 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in h*nmol/L.
Part 2 (DC): Cmax,4768,SS: maximum observed plasma concentration of NNC0113-4768 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 50, 78 and 106
  Measured in nmol/L.
Part 3 Japanese (JP): AUCτ,sema,SS: area under the semaglutide plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in h*nmol/L.
Part 3 (JP): Cmax,sema,SS: maximum observed plasma concentration of semaglutide at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nmol/L.
Part 3 (JP): AUCτ,6856,SS: area under the NNC0113-6856 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in h*nmol/L.
Part 3 (JP): Cmax,6856,SS: maximum observed plasma concentration of NNC0113-6856 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nmol/L.
Part 3 (JP): AUCτ,4768,SS: area under the NNC0113-4768 plasma concentration-time curve during a dosing interval τ at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in h*nmol/L.
Part 3 (JP): Cmax,4768,SS: maximum observed plasma concentration of NNC0113-4768 at steady state | From 0 to 168 hours after fourth dosing with the same dose at days 22, 50, 78 and 106
  Measured in nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com